CLINICAL TRIAL: NCT02808767
Title: Comparison of Prasugrel and Ticagrelor in the Treatment of Acute Myocardial Infarction
Acronym: PRAGUE-18
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Zuzana Motovska, Accociate Professor, Faculty Hospital Kralovske Vinohrady
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK-VP/04/2013
Record Dates: First submitted 2016-06-12; First posted 2016-06-22 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Myocardial Infarction; Angioplasty, Balloon, Coronary; Platelet Aggregation Inhibitors
Keywords: Acute myocardial infarction; Primary coronary intervention; Antiplatelet therapy
MeSH Terms: conditions — Myocardial Infarction | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients treated with Prasugrel (Experimental): Prasugrel Loading dose: 60 mg Maintenance dose: 10 mg once-daily; patients >75 years of age or < 60 kg of weight receive a maintenance dose of 5 mg o.d.
  Interventions: Drug: Prasugrel
- Patients treated with ticagrelor (Experimental): Ticagrelor Loading dose: 180 mg Maintenance dose: 90mg twice-daily
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 60 mg loading dose and 10mg/5mg once daily maintenance dose
  Other Names: Efient
  Arms: Patients treated with Prasugrel
Drug: Ticagrelor — Ticagrelor 180 mg loading dose and 90 mg twice daily maintenance dose
  Other Names: Brilique
  Arms: Patients treated with ticagrelor

SUMMARY:
This study evaluates the efficacy of Prasugrel and Ticagrelor in the treatment of acute myocardial infarction.

DETAILED DESCRIPTION:
Study objectives:

1. Compare the efficacy and safety of prasugrel and ticagrelor in acute myocardial infarction treated with emergent PCI.
2. Assess the safety of switching to clopidogrel after remission of the acute phase of MI in patients for whom economic barriers do not allow to continue treatment with prasugrel or ticagrelor. All randomized patients with acute myocardial infarction have been treated with standard therapeutic procedures in accordance with the guidelines of European Society of Cardiology (ESC). Participation of patients in the study is not connected to any deviations from the ESC guidelines recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myocardial infarction (> 1mm ST elevation in at least 2 related leads or ST depression > 2mm in 3 leads or new BBB) with an indication to emergent (within 120 minut from admission to the PCI center) coronary angiography and PCI,
2. Signed informed consent.

Exclusion Criteria:

1. History of stroke,
2. Serious bleeding within last 6 months,
3. Indication to an oral anticoagulation (e.g. atrial fibrillation, artificial valve, thromboembolism etc...)
4. Use of ≥ 300 mg of clopidogrel or another antiplatelet agent (except of aspirin and lower dose of clopidogrel) before randomization,
5. Low body weight (<60 kg) in an older patient (>75 years of age),
6. Moderate or severe liver dysfunction,
7. Ongoing therapy with a strong CYP3A4 inhibitor (e.g. ketoconazole, clarythromycine, nefazodone, ritonavir, atazanavit),
8. Hypersensitivity to prasugrel or ticagrelor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1226 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Composite primary outcome measure consisting of Death / Re-infarction / Stroke / Serious bleeding requiring transfusion or prolonged hospitalization / Urgent Target Vessel Revascularization. | Within 7 days after Randomization.
  Definitions:
  Death defined as summary of death from any cause. Re-infarcion defined according to the Third Universal Definition of Myocardial Infarction.
  Stroke defined as the rapid onset of new neurological deficit caused by an ischemic or hemorrhagic central nervous system event with symptoms that lasted at least 24 hours after onset or leading to death.
  Urgent Target Vessel Revascularization defined as a new emergent/urgent revascularization of the vessel dilated at the initial procedure driven by recurrent signs of ischemia occurring after completion of initial PCI.
  Units: The percentage of randomized patients is the total number of randomized patients experiencing Death / Re-infarction / Stroke / Serious bleeding requiring transfusion or prolonged hospitalization / Urgent Target Vessel Revascularization divided by number of randomized patients in the treatment arm multiplied by 100.
  Primary endpoint is adjudicated by the Independent Control committee

SECONDARY OUTCOMES:
Composite secondary outcome measure consisting of Cadiovascular death / Non-fatal myocardial infarction / Stroke. | Within 30 days and one year after Randomization.
  Definition:
  Cardiovascular death defined as a death with a demonstrable cardiovascular cause, or any death that is not clearly attributable to a non-cardiovascular cause.
  Non-fatal myocardial infarction must be distinct from the index event and is defined according to the Third Universal Definition of Myocardial Infarction.
  Units: The percentage of randomized patients is the total number of randomized patients experiencing Cadiovascular death / Non-fatal myocardial infarction / Stroke divided by number of randomized patients in the treatment arm multiplied by 100.
Stent thrombosis. | Within 30 days and one year after Randomization.
  Definition: Academic Research Consortium (ARC) criteria were used to define ST. Units: The percentage of randomized patients is the total number of randomized patients experiencing Stent thrombosis divided by number of randomized patients in the treatment arm multiplied by 100.
Occurence of bleeding according to the TIMI and BARC criteria. | Within 30 days and one year after Randomization.
  TIMI criteria - Thrombolysis In Myocardial Infarction Criteria BARC criteria - Bleeding Academic Research Consortium criteria Units: The percentage of randomized patients is the total number of randomized patients experiencing bleeding according to the TIMI and BARC criteria divided by number of randomized patients in the treatment arm multiplied by 100.

OTHER OUTCOMES:
Composite outcome measure consisting of Cadiovascular death / Non-fatal myocardial infarction / Stroke in patients with Killip III/IV. | Within 7 days after Randomization.
  The percentage of randomized patients is the total number of randomized patients with Killip class III or IV experiencing Cardiovascular death / Non-fatal myocardial infarction / Stroke divided by number of randomized patients with Killip class III or IV in the treatment arm multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Motovska, MD PhD, Principal Investigator — University Hospital Kralovske Vinohrady, Prague, Czech Republic; Petr Widimsky, Prof MD DrSc, Principal Investigator — University Hospital Kralovske Vinohrady, Prague, Czech Republic
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Motovska Z, Hlinomaz O, Miklik R, Hromadka M, Varvarovsky I, Dusek J, Knot J, Jarkovsky J, Kala P, Rokyta R, Tousek F, Kramarikova P, Majtan B, Simek S, Branny M, Mrozek J, Cervinka P, Ostransky J, Widimsky P; PRAGUE-18 Study Group. Prasugrel Versus Ticagrelor in Patients With Acute Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention: Multicenter Randomized PRAGUE-18 Study. Circulation. 2016 Nov 22;134(21):1603-1612. doi: 10.1161/CIRCULATIONAHA.116.024823. Epub 2016 Aug 30. PMID 27576777
- [Derived] Motovska Z, Hlinomaz O, Kala P, Hromadka M, Knot J, Varvarovsky I, Dusek J, Jarkovsky J, Miklik R, Rokyta R, Tousek F, Kramarikova P, Svoboda M, Majtan B, Simek S, Branny M, Mrozek J, Cervinka P, Ostransky J, Widimsky P; PRAGUE-18 Study Group. 1-Year Outcomes of Patients Undergoing Primary Angioplasty for Myocardial Infarction Treated With Prasugrel Versus Ticagrelor. J Am Coll Cardiol. 2018 Jan 30;71(4):371-381. doi: 10.1016/j.jacc.2017.11.008. Epub 2017 Nov 14. PMID 29154813